CLINICAL TRIAL: NCT03683095
Title: Efficacy of Lymphovenous Bypass in the Treatment of Extremity Lymphedema
Status: Withdrawn | Type: Observational
Why Stopped: Insufficient resources
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 20180289-01H
Record Dates: First submitted 2018-09-16; First posted 2018-09-25 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Lymph Leakage
Keywords: Lymphedema; Lymphovenous bypass
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lymphovenous bypass: Patients with extremity lymphedema treated with lymphovenous bypass.
  Interventions: Procedure: Lymphovenous bypass

INTERVENTIONS:
Procedure: Lymphovenous bypass — Lymphovenous bypass will be performed under general anesthetic. Indocyanine green lymphangiography will be performed by injecting indocyanine green into each finger / toe web of the lymphedematous limb and mapping the lymphatic system with the NOVADAQ SPY Fluorescence Imaging (Mississauga, Canada).
  Subdermal dissection of lymphatics and venules will be carried out under a surgical microscope. Lymphatic vessels will be anastomosed to adjacent recipient venules to create the bypass between the lymphatic and the venous systems. In total, 1-5 anastomoses will be performed. This will require 1-5 incisions, each with a length of 2-3 cm.
  Postoperatively, the limb will be wrapped loosely with compression bandages. No special postoperative monitoring is required.
  The surgery will be performed on an outpatient basis with no planned hospital stay.

SUMMARY:
BACKGROUND: Lymphedema is a pathologic soft tissue swelling that arises secondary to disruption of the lymphatic system. Lymphedema affects approximately 250 million people worldwide and causes significant physical and psychological morbidity. There is no definitive treatment for lymphedema. Lymphovenous bypass - microsurgically anastomosing lymphatic channels and venules - has demonstrated promising results in the treatment of lymphedema. PURPOSE: The purpose of this study is to determine the efficacy of lymphovenous bypass in treating extremity lymphedema. METHODS: This is a prospective, single-arm, cohort study. Eligible patients between 18-70 years of age with extremity lymphedema will undergo lymphovenous bypass. The primary outcome measure will be extremity volume and the secondary outcome measure will be quality of life assessed by a validated assessment tool for lymphedema of the limbs (LYMQOL). Patients will be assessed preoperatively and at 3, 6, 9, and 12-months postoperatively. Each participant will serve as their own control.

Primary and secondary outcome measures will be assessed with paired t-tests. With a sample size of 9 patients we will have at least 80% power to reject the null hypothesis assuming an alpha level of 0.01. To further increase the power and to account for patients lost to follow-up the investigators will target a patient recruitment of 20.

The findings of this study will help further elucidate the role of lymphovenous bypass in the treatment of extremity lymphedema.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years.
2. Lymphedema of the upper or lower extremity.
3. International Society of Lymphology Stage I-II.

Exclusion Criteria:

1. Significant comorbidities that would preclude a patient from receiving a general anesthetic.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (18-70 years) with International Society of Lymphology Stage I-II lymphedema of the upper or lower extremity will be eligible for lymphovenous bypass.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Extremity volume (v) | Assessed preoperatively and 12-months postoperatively.
  Extremity volume will be calculated using the truncated cone formula based on limb circumference measurements.

SECONDARY OUTCOMES:
Quality of life assessment tool for lymphedema of the limbs (LYMQOL). | Assessed preoperatively and 12-months postoperatively.
  Quality of life assessment tool for lymphedema of the limbs.

OTHER OUTCOMES:
Number of episodes of cellulitis (n / year) | Patient estimate from the 12-months preoperatively compared with 12-months postoperatively.
  Number of episodes of cellulitis requiring antimicrobial therapy (n / year).
Need for ongoing compression therapy (yes / no) | Assessed preoperatively and 12-months postoperatively.
  Need for ongoing compression therapy as defined by the use of acute bandaging, compression garments, or manual compression therapy (yes / no).

CONTACTS AND LOCATIONS:
Overall Officials: Moein Momtazi, MD, Principal Investigator — Division of Plastic & Reconstructive Surgery, Department of Surgery, University of Ottawa

IPD SHARING:
Plan to Share IPD: No